CLINICAL TRIAL: NCT06480903
Title: Exploratory Study of Plasma Epstein Barr Virus (EBV) DNA Clearance During Proton Beam Therapy (PBT) for Nasopharyngeal Carcinoma (NPC)
Brief Title: Exploratory Study of EBV DNA Titre Clearance Whilst on Proton Beam Therapy
Acronym: ClearED
Status: Not yet recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp237
Record Dates: First submitted 2024-06-18; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Nasopharyngeal Carcinoma; Head and Neck Cancer; Nasopharyngeal Cancer; Epstein-Barr Virus
Keywords: Nasopharyngeal, cancer, proton beam, epstein-barr virus
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Head and Neck Neoplasms; Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Epstein-barr virus DNA, within blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
How does plasma Epstein-Barr Virus (EBV) DNA level change during definitive radiation therapy for nasopharyngeal carcinoma (NPC) in the teenage and young adult cohort and does it correlate with outcomes?

DETAILED DESCRIPTION:
Children with NPC achieve superior survival outcomes compared to adults (10) and the prognostic value of plasma Epstein-Barr Virus (EBV) DNA has not been studied in children. Integration of MRI into early treatment response assessment will add further prognostic value and permits response-adapted therapy which can improve quality of survivorship children through toxicity reduction. It also allows identification of patients who either have had or are likely to have a suboptimal response to treatment, facilitating the potential consideration of treatment escalation.

The sample size of this study is not intended to change clinical practice, but rather provide a basis for international collaboration to achieve larger patient numbers.

ELIGIBILITY:
Inclusion Criteria:

* Children and young adults (8-30 years old)
* Pathologically confirmed EBV-positive nasopharyngeal carcinoma
* Stage I-IVA (AJCC 8th Edition)
* Planned to commence curative-intent radiation therapy

Exclusion Criteria:

* Recurrent NPC
* Concurrent or previously treated EBV-associated malignancy
* Prior radiation therapy
* Contraindications to MRI
* General anaesthetic requirement for MRI

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, teenagers and young adults with nasopharyngeal carcinoma (age 8-30 years old)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Plasma EBV during proton beam RT | 6 weeks
  Taken weekly, prior to each session of chemotherapy. Change in plasma EBV DNA levels (EBV VCA-IgM Ab) from each blood sample time point.

SECONDARY OUTCOMES:
EBV and tumour correlates | 2 years
  Taken weekly, prior to each session of chemotherapy. Change in plasma EBV DNA levels (EBV VCA-IgM Ab) from each blood sample. Assessment whether EBV plasma clearance predicts tumour response.

IPD SHARING:
Plan to Share IPD: No
Aggregated data only

REFERENCES:
- [Background] Twu CW, Wang WY, Liang WM, Jan JS, Jiang RS, Chao J, Jin YT, Lin JC. Comparison of the prognostic impact of serum anti-EBV antibody and plasma EBV DNA assays in nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2007 Jan 1;67(1):130-7. doi: 10.1016/j.ijrobp.2006.07.012. Epub 2006 Sep 18. PMID 16979842
- [Background] Chan AT, Lo YM, Zee B, Chan LY, Ma BB, Leung SF, Mo F, Lai M, Ho S, Huang DP, Johnson PJ. Plasma Epstein-Barr virus DNA and residual disease after radiotherapy for undifferentiated nasopharyngeal carcinoma. J Natl Cancer Inst. 2002 Nov 6;94(21):1614-9. doi: 10.1093/jnci/94.21.1614. PMID 12419787
- [Background] Chan SK, Chan SY, Choi HC, Tong CC, Lam KO, Kwong DL, Vardhanabhuti V, Leung TW, Luk MY, Lee AW, Lee VH. Prognostication of Half-Life Clearance of Plasma EBV DNA in Previously Untreated Non-metastatic Nasopharyngeal Carcinoma Treated With Radical Intensity-Modulated Radiation Therapy. Front Oncol. 2020 Aug 21;10:1417. doi: 10.3389/fonc.2020.01417. eCollection 2020. PMID 32974150